CLINICAL TRIAL: NCT03112915
Title: Comparison of Quadratus Lumborum Block and Transversus Abdominis Plane Block for Postoperative Pain Control After Laparoscopic Cholecystectomy
Brief Title: Comparison of the Quadratus Lumborum Block With the Transversus Abdominis Plan Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Merve Kacan, Assistant doctor, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2017-02-27; First posted 2017-04-13 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; Laparoscopic cholecystectomy; Quadratus lumborum block; transversus abdominis plan block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trail
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind randomized controlled trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB: Quadratus lumborum block (Active Comparator): QLB: Quadratus lumborum block :Quadratus Lumborum block group (QL)
  patients will receive a bilateral Quadratus Lumborum block using Bupivicaine 0.25 %
  Interventions: Procedure: quadratus lumborum block
- TAP: transversus abdominis plan block (Active Comparator): TAP: Transversus abdominis plane block (TAP)
  patients will receive a bilateral TAP block using Bupivicaine 0.25%
  Interventions: Procedure: Transversus abdominis plan block

INTERVENTIONS:
Procedure: quadratus lumborum block — QLB: Quadratus lumborum block : 20 mL of 0.25% bupivacaine will be administered between the quadratus lumborum and the psoas major muscle bilaterally in the lateral decubitus position
  Other Names: QLB
  Arms: QLB: Quadratus lumborum block
Procedure: Transversus abdominis plan block — TAP: transversus abdominis plan block: 20 mL of 0.25% bupivacaine will be administered between the internal oblique muscle and the transversus abdominis muscle bilaterally in the supine position
  Other Names: TAP block
  Arms: TAP: transversus abdominis plan block

SUMMARY:
In this study, investigators aimed to compare the Quadratus Lumborum Block and the Transversus Abdominis Plan Block for postoperative pain control after laparoscopic cholecystectomy

DETAILED DESCRIPTION:
After ethical committee approval, informed written consent will be obtained from all patients.

A Sample size of 60 patients (30 per group) was calculated based on 15% reduction in morphine consumption with 0.05% significance and a power of 0.8.

Consenting patients scheduled to have elective laparoscopic cholecystectomy under general anesthesia will be randomized to receive bilateral QLB or TAP before the surgery. The dose of local anesthetic in both groups will be 20 ml 0.25% Bupivacaine. Allocation to either group will be done using permuted block randomization method.

Patients will be taken to the block room 1 hour before surgery. ECG, NIBP and SpO2 monitor will be done. The IV access route will be provided. The patient will be given 0.03 mg / kg IV midazolam for routine premedication. Block will be applied by a blind anesthetist to the other data of the study. Under ultrasound guidance a 22 Gauge Sonoplex needle will be used for both techniques. The calculated dose of local anesthetic will be injected bilaterally with intermittent aspiration. The spread of injectate will be seed on ultrasound.

The procedure time for both blocks will be recorded and 30 minutes after the procedure is completed, and the patient will be taken to the operation room. General anesthesia will be applied to the patient in the operation procedure in the standard procedure. Intraoperative heart rate and / or mean arterial pressure is increased to 20% of the basal value and 0.5 mcg / kg IV fentanyl will be added. 30 minutes before the end of operation, 1 mg IV paracetamol and NSAID (dexketoprofen) 50 mg IV will be administered to the patient before extubation. The patient will be infected with IV PCA in the morphine. PC 1 mg IV bolus dose will be adjusted to 10 minutes of locked-out period. In the postoperative period, 4 * 1 gr / 24 h IV paracetamol will be given to each patient.

All patients will be assessed postoperatively by a blinded investigator: in the post-anesthesia care unit and at 0, 2, 4, 6, 12 and 24 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3
* elective Laparoscopic cholecystectomy
* 19-65 years
* Written informed consent

Exclusion Criteria:

* Patient refusal Local infection at the site of injection
* Allergy to study medications Sepsis Anatomic abnormalities Systemic anticoagulation or coagulopathy - Inability to comprehend or participate in pain scoring system
* Inability to use intravenous patient controlled analgesia

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-09-12 (Estimated)

PRIMARY OUTCOMES:
Total cumulative morphine consumption | 24 hour
  Total cumulative morphine dose in mg used in the first 24 hours after surgery

SECONDARY OUTCOMES:
Severity of postoperative pain via visual analogue pain scale (VAS) | 24 hour
  VAS range from 0 for no pain to 10 for worst pain imaginable
Nausea or vomiting | 24 hour
  0 = No Nausea
  1. = Mild Nausea.
  2. = Moderate 3 = Severe Nausea or Vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Kecioren ETH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28154824
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27755488